CLINICAL TRIAL: NCT05612464
Title: Enhancing Cortical Sensorimotor Processing in Children/Young People With Dystonia and Dystonic Cerebral Palsy - An Observational Study to Evaluate Whether Neurofeedback Can Enhance Modulation of the mu Brain Rhythm in Children and Young People With Dystonia/Dystonic Cerebral Palsy
Brief Title: Enhancing Sensorimotor Processing in Children With Dystonia
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); Imperial College London (Other); University of Bristol (Other); University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: 317454
Record Dates: First submitted 2022-10-24; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Dystonia; Dystonic Cerebral Palsy; Dystonia, Secondary; Dystonia, Primary; Dystonia; Idiopathic
MeSH Terms: conditions — Dystonia; Dystonic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary dystonia group (genetic or idiopathic)
  Interventions: Other: No intervention
- Dystonic cerebral palsy group
  Interventions: Other: No intervention
- Control group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Dystonia is a severely disabling movement disorder with no cure, in which people suffer painful muscle spasms causing twisting movements and abnormal postures. There are many causes, including genetic conditions and brain injury. The most common cause in childhood is dystonic cerebral palsy (CP) which often affects the whole body.

The underlying mechanisms are unknown, but there is growing evidence to implicate abnormal brain processing by the brain of incoming "sensory" information (e.g., signals to the brain from our senses of touch and body position): the distorted perception of these signals disrupts the way the brain produces instructions for planning and performing movements.

The investigator's previous studies have shown that the way the brain processes sensory information related to movement is abnormal in children with dystonia and dystonic CP, by using methods that record the EEG (electroencephalogram - brain wave signals) and/or EMG (electromyogram - electrical signal from muscles). A specific brain rhythm (called mu) typically shows well-defined changes in response to movement, and reflects processing of sensory information. The investigator's work shows these rhythm changes are abnormal in children with dystonia/dystonic CP.

This study will explore if these findings can improve treatment. In particular the study team will investigate whether children and young people with dystonia/dystonic CP can enhance these mu rhythm responses during a movement task by using feedback of their brain rhythms displayed as a cartoon/game on a computer. The investigators will also assess whether enhanced mu activity is associated with improved movement control. This would open future possibilities to use such devices for therapy/rehabilitation.

Children and young people with dystonia/dystonic CP aged 5-25 years will be recruited, along with age-matched controls. Studies will last 2-3 hours with time for breaks and will be conducted at Evelina London Children's Hospital and Barts Health Trust, with the option for home visits if preferable for families.

ELIGIBILITY:
Key inclusion criteria

Control Group:

* Age 5 -25 years
* No known disorder of movement
* Able to understand and participate in study.

Primary dystonia group (isolated genetic or idiopathic):

* Age 5-25 years
* Clinical dystonia - as confirmed on clinical assessment by consultant paediatric neurologist.
* Genetic or idiopathic aetiology.
* No other neurological abnormality.
* Normal cranial magnetic resonance imaging (MRI).
* Able to understand and participate in study.

Dystonic Cerebral Palsy Group:

* Age 5-25 years
* Clinical dystonia/dyskinesia - as confirmed on clinical assessment by consultant paediatric neurologist.
* Documented history of perinatal hypoxic-ischaemic encephalopathy (HIE), prematurity <35 weeks or kernicterus.
* Predominant dystonia/dyskinesia / Minimal spasticity
* MRI findings in keeping with acute perinatal HIE, prematurity or kernicterus (including classical pattern of damage to thalami, basal ganglia and peri-rolandic cortex, periventricular leukomalacia or ischaemic parenchymal injury).
* Able to understand and participate in study.

Key exclusion criteria

Control Group:

* Age <5 or >25 years
* Any known disorder of movement.

Primary dystonia group (isolated genetic or idiopathic):

* Age < 5 or >25 years
* Presence of other neurological abnormality in addition to dystonia.
* Abnormal cranial MRI.

Dystonic Cerebral Palsy Group:

* Age < 5 or >25 years
* No clear history of perinatal HIE, prematurity or kernicterus.
* Predominant spasticity.
* MRI scan not compatible with perinatal HIE, prematurity or kernicterus

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Population to be researched is children/young people with dystonia / dystonic cerebral palsy.
  Age range 5-25 years
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in mu modulation between trials with and without biofeedback | During the procedure

IPD SHARING:
Plan to Share IPD: Yes
The research team will have exclusive use of the data for the project duration and five years afterwards to allow for publications to be achieved. After this period, the majority of data would be made available for data sharing via the King's College London data repository. Only non-identifiable data will be available.
Supporting Information: Study Protocol
Time Frame: Data will be available approximately 5 years after the end of the study
Access Criteria: The data would be deposited within the institutional data repository at King's College London (KCL). Each dataset will have a data sharing policy, in line with MRC (Medical Research Council) guidance and KCL policies. Governance of access will be in line with these study-specific policies. The PI will be involved in making the decision-making process for access requests, along with the repository team.